CLINICAL TRIAL: NCT02364479
Title: Treatment of Active Axial Spondyloarthritis by Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ IgG Fc Fusion Protein Injection: a Randomized, Double-blind, Multicentral Clinical Trial to Investigate the Efficacy and Safety of Yisaipu®
Brief Title: Treatment of Axial Spondyloarthritis by Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ IgG Fc Fusion Protein
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gu Jieruo, Division of Rheumatology of Third Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: [2013]2-21
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Spondyloarthritis
Keywords: relapse; Yisaipu
MeSH Terms: conditions — Spondylarthritis; Recurrence | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 50mg etanercept (Experimental): Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ IgG Fc Fusion Protein Injection, 50mg per week, Subcutaneous injection
  Interventions: Drug: 50mg Yisaipu
- 25mg etanercept (Experimental): Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ IgG Fc Fusion Protein Injectio, 25mg per week, Subcutaneous injection
  Interventions: Drug: 25mg etanercept
- Placebo (Placebo Comparator): Placebo, Subcutaneous injection per week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 50mg Yisaipu — Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ IgG Fc Fusion Protein Injection, 50mg per week
  Other Names: 50mg entanercept(Yisaipu)
  Arms: 50mg etanercept
Drug: 25mg etanercept — Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ IgG Fc Fusion Protein Injection, 25mg per week
  Other Names: 25mg entanercept(Yisaipu)
  Arms: 25mg etanercept
Drug: Placebo — The injection method and frequency of placebo is the same as the other arms.
  Other Names: placebo arm
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, multicentral clinical trial to investigate the efficacy and safety of Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ IgG Fc fusion protein injection (Yisaipu®) in the treatment of active axial spondyloarthritis(SpA). The primary purpose is to assess the different situations in maintaining treatment programme in SpA patients with controlled inflammation by Yisaipu®. And the second purpose is to assess the eficacy and safety of Yisaipu® in axial SpAs. The trial will include 150 patients with stable NSAIDs therapy, and at the first stage they will receive 24-week full-dose of Yisaipu®. Then at the second stage the patients who achieve low disease activity (LDA, ASDAS<2.1) at 24th week will be randomizedly divided into three group: full-dose of Yisaipu® group, half-dose of Yisaipu® group and placebo group. And the blind stage will last for 48 weeks. Patients who complete the 72-week therapy or achieve disease-flare criteria during the blind stage would finish the study.

DETAILED DESCRIPTION:
This randomised controlled trial enrolled adult patients aged 18 years or older diagnosed with non-radiographic axial spondyloarthritis at 3 centres in China. Patients had to fulfil ASAS axial spondyloarthritis criteria but could not fulfil the modified New York radiologic criterion for ankylosing spondylitis,and had to have objective evidence of active inflammation or chronic structral change，such as bone erosion or fat metaplasia in the sacroiliac joints on MRI at screening. Active disease activity was defined as a disease activity score in ASDAS-CRP ≥2.1,or Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] ≥4 on a numerical rating scale of 0-10, and an inadequate response to more than one non-steroidal anti-inflammatory drugs (NSAIDs) for 4 weeks at least, intolerance to NSAIDs, or contraindication for NSAIDs. No change in NSAIDs dose was required from 2 weeks before screening to the end of the study. Dose stability or discontinuation was required for 4 weeks before baseline for concomitant DMARDs or corticosteroids (prednisone or equivalent at a dose of less than 10 mg/day). Chinese herbal medicine, physical therapy, or live (attenuated) vaccine, or intravenous immunoglobulin IgG, was required for discontinuation and wash period for at least 4 weeks. Patients were excluded if they had previously taken or were taking biologic treatment, any biologic Dmards such as IL-6 or CD-20 inhibitors. Patients with latent tuberculosis infection were included only when local guidelines were followed for prophylactic treatment and if treatment was initiated before Yisaipu.

All patients provided written informed consent, and the study protocol was approved by an institutional review board or independent ethics committee at each study site. The study was conducted in accordance with applicable regulations and the ethical principles of Good Clinical Practice as defined by the International Conference on Harmonisation (ICH) and the Declaration of Helsinki.

A randomized envelope was used to enrol all patients at the baseline visit and to randomly assign qualifying patients in a 1:1:1 ratio to receive either blinded Yisaipu 50 mg subcutaneously every week or 25 mg subcutaneously every week or matching placebo at week 24. All study personnel, including the sponsor (with the exception of the Sanshengguojian drug supply management team), investigator, and study site personnel, and the patient remained blinded to treatment throughout the double-blinded period from week 24 through week 72 of the study. Investigational products were provided to maintain blinding.

In the initial open-label period, enrolled patients were given subcutaneous injections of 50 mg Yisaipu every week for 36 weeks. Participants were given the dose of NSAIDs they had been receiving at screening; a dose decrease or discontinuation was allowed when the patients were intolerance to NSAIDs, or contraindication for NSAIDs. Patients who achieved clinical remission, defined as achieving ASDAS inactive or moderate disease (ASDAS score <2.1) at weeks 24, were randomly assigned to receive either blinded 50mg Yisaipu (continuation arm), 25mg Yisaipu(reduction arm) or matching placebo (withdrawal arm) for 48 weeks during the double-blind period, for a total of 72 weeks of treatment.

During the double-blind period, patients who experienced a flare (defined as an increase in BASDAI ≥2 points compare to the BASDAI score when randomization) were allocate to termination of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the 2009 ASAS criteria for axial spondyloarthritis(SpA), and without bilateral more than grave 2 or unilateral more than grave 3 sacroilitis on X ray plan
* Active disease phase of SpA, defined as BASDAI≥4 or ASDAS≥2.1
* Inadequate response to NSAID≥4 week
* Application of NSAID with stable dose for no less than 2 weeks
* Stable dose of prenisone for at least four weeks at ≤10mg per day if used at screening, or stop use for at least 4 weeks.
* Stable dose of any DMARD for at least four weeks if used at screening, or stop use for at least 4 weeks
* Stop and receiving washing out for at least 4 week if receiving Chinese traditional drug for AS, physical treatment, vaccication or IVIG.
* The lab exam should achieve the criteria as below: Hb≥85g/L, 3.5×109/L≤WBC count≤10×109/L, PLT≥ lower limit of normal range, ALT≤2 fold of upper limit of normal range, serum creatine ≤upper limit of normal range.
* Negative pregnacy test for female patients. And promise to carry out contraception during the trial and 6 weeks after the trial is ended.
* Sign the informed consent.

Exclusion criteria:

* Previous application of any biologic agents.
* Allergic to any element of Yisaipu®
* Intolerance to NASID.
* History of active tubercolosis, or radiographic evidence of present or previous history of pulmonary tubercolosis, or close contact with patients with tubercolosis, or with high risk of infection of tubercolosis such as immune suppression status, or strong positive of PPD skin test with diameter ≥10mm.
* Presence of acute infection or acute onset of chronic infection at screen.
* Invasive fungal infection or conditional infection within 6 months prior to screen.
* Present or history of serious liver disease.
* History of infection on artifitial joints.
* Organ transplantation surgery within 6 months prior to screen.
* Presence of other autoimmune diseases, including IBD, psoriasis, uveitis, SLE, multiple sclerosis, etc.
* History of congestive heart failure.
* History of malignancies within 5 years prior to screen, excluding complete resection of squamous cell carcinoma, or basal cell carcinoma or cervical carcinoma in situ.
* AIDS or HIV infection.
* History of lymphoma or lymphoproliferative disorders.
* Presence of serious disorder of important organs or system.
* Presence of factors which may influence the compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-08-28 (Actual)

PRIMARY OUTCOMES:
proportion of patients achieving ASDAS<2.1 | 72 week
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period

SECONDARY OUTCOMES:
proportion of patients achieving ASDAS<1.3 | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
proportion of ASDAS major improvement | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
proportion of ASDAS clinically important improvement | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
ASAS 20 | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
ASAS 40 | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
ASAS5/6 | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
ASAS PR | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
BASDAI50 | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
BASDAI | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
BASFI | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
BASMI | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
spinal pain score | 72 weeks
  The unabbreviated scale title is VAS from 0 to 100mm. 100 mm mean the most severe pain
patient global assessment(PGA) score | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
physician global assessment(PhGA) score | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
ESR | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period
CRP | 72 weeks
  in the groups given 50 mg Yisaipu, 25mg Yisaipu compared to placebo in the double-blind period

CONTACTS AND LOCATIONS:
Overall Officials: Jieruo Gu, Professor, Principal Investigator — 3rd Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Department of Rheumatology, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China